CLINICAL TRIAL: NCT04448808
Title: Treating Nightmares in Posttraumatic Stress Disorder With Dronabinol: A Randomized Controlled Study (THC PTSD-trial)
Brief Title: Treating Nightmares in Posttraumatic Stress Disorder With Dronabinol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Bionorica SE (Industry)
Responsible Party: Principal Investigator, Stefan Roepke, Prof. Dr. Stefan Roepke, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THC-PTBS
Record Dates: First submitted 2020-06-16; First posted 2020-06-26 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Nightmares; Posttraumatic Stress Disorder; Dronabinol
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Randomized controlled study (double-blind)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BX-1 (dronabinol) (Experimental): BX-1
  Interventions: Drug: BX-1
- Placebo (Placebo Comparator): Placebo of BX-1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BX-1 — BX-1 (dronabinol), oral solution. All patients enrolled establish their individually tolerable dose by dose Titration.
  Arms: BX-1 (dronabinol)
Drug: Placebo — Placebo of BX-1, oral solution
  Arms: Placebo

SUMMARY:
This randomized controlled exploratory phase II trial will test the hypothesis that oral dronabinol improves nightmares (primary outcome) and other PTSD symptoms (secondary outcomes) to a greater extent than placebo over a ten week intervention phase in a parallel group design.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of posttraumatic stress disorder (PTSD) according to DSM 5 with a 20 item CAPS-5 total score ≥ 26
2. At least two nightmares a week, an intensity score ≥ 2, with a CAPS-IV B2 (frequency and intensity for the last week) score ≥ 5
3. Men and women between 18 and 65 years of age
4. Written informed consent
5. The patient has the capacity to give consent (He/she is able to understand the nature and anticipated effects/side effects of the proposed medical intervention)
6. The patient is not breastfeeding
7. Women of child-bearing potential must have a negative urine or serum pregnancy test
8. All participants must use highly effective contraception
9. The patient received stable pharmacological medication for at least 4 weeks prior to study entry (any changes in medication dose or frequency of therapy must be answered with no)

Exclusion Criteria:

1. Lifetime cannabis use disorder
2. Current substance/alcohol use disorder (≤ 3 months);
3. Acute suicidality;
4. Psychotic disorder;
5. Bipolar disorder;
6. Current anorexia nervosa;
7. Current major depressive episodes and a MADRS score > 29;
8. Dementia;
9. Trauma-focused psychotherapy four weeks before the trial
10. Initiation of sleep medication 4 weeks prior screening or initiation of alpha adrenergic agents 4 weeks prior to screening
11. Acute or unstable medical illness.
12. Epilepsy
13. Relevant heart diseases
14. Known HIV- and/or active Hepatitis-B- or Hepatitis-C-infection
15. Current or past malignant illness
16. The patient is unwilling to consent to saving, processing and propagation of pseudonymized medical data for study reasons
17. Patients, who may be dependent on the sponsor, the investigator or the trial sites, have to be excluded from the trial
18. The patient is legally detained in an official institution
19. The patient does have a known allergy or contraindication against Dronabinol
20. The patient does have clinically significant abnormalities in 12-lead ECG
21. The patient does have clinically significant laboratory abnormalities
22. The patient did participate in other interventional trials during the 3 months before and at the time of this trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Frequency and intensity of nightmares | 10 weeks
  Frequency and intensity of nightmares, measured with the Clinician-Administered PTSD Scale-IV (CAPS-IV) B2 score for the last week, range 0-8. A lower score indicates less frequent and/or intense nightmares.

SECONDARY OUTCOMES:
Change from baseline of the frequency and intensity of nightmares | 1, 2, 3, 4,6 and 8 weeks
  Change from baseline of the frequency and intensity of nightmares, measured with the Clinician-Administered PTSD Scale-IV (CAPS-IV) B2 score for the last week, range 0-8.
Change from baseline of the CAPS-5 total score | 6 and 10 weeks
  Change from baseline of the CAPS-5 total score (overall PTSD symptoms, last week)
Change from baseline of the Pittsburgh Sleep Quality Index-Addendum for PTSD | 6 and 10 weeks
  Change from baseline of the Pittsburgh Sleep Quality Index-Addendum for PTSD (PSQI A) (PTSD related sleep symptoms)
Change from baseline of the Montgomery-Åsberg Depression Rating Scale | 4 and 10 weeks
  Change from baseline of the Montgomery-Åsberg Depression Rating Scale (MADRS, depressive symptoms)
Weekly mean of change from baseline of daily total sleep time | during 10 weeks
  Weekly mean of change from baseline of the patients daily total sleep time (in minutes), assessed with sleep diaries
Weekly mean of change from baseline of the patients sleep onset latency at night | during 10 weeks
  Weekly mean of change from baseline of the patients sleep onset latency at night (in minutes), assessed with sleep diaries
Weekly mean of change from baseline of the patients recuperation of night sleep | during 10 weeks
  Weekly mean of change from baseline of the patients recuperation of night sleep (5-point Likert scale, 1 = very much; 5 = not at all), assessed with sleep diaries
Weekly mean of change from baseline of the patients time awake at night | during 10 weeks
  Weekly mean of change from baseline of the patients time awake at night (in minutes), assessed with sleep diaries
Weekly mean of change from baseline of the patients number of nightmares last night | during 10 weeks
  Weekly mean of change from baseline of the patients number of nightmares last night (0, 1, 3, 4 or more) assessed with sleep diaries
Weekly mean of change from baseline of the patients intensity of nightmares | during 10 weeks
  Weekly mean of change from baseline of the patients intensity of nightmares (5-point Likert scale, 0 = not at all; 5 = extreme) assessed with sleep diaries
Change from baseline of PTSD symptoms assessed with the PTSD Checklist for DSM-5 | 6 and 10 weeks
  Change from baseline of PTSD symptoms assessed with the PTSD Checklist for DSM-5 (PCL-5)
Change from baseline of the Borderline Symptom List 23 | 6 and 10 weeks
  Change from baseline of the Borderline Symptom List 23 (BSL-23) score
Change from baseline of the Health-Related Quality of Life | 6 and 10 weeks
  Change from baseline of the Health-Related Quality of Life (EQ-5D) score
Overall patients status measured by the Patient Global Impression of Change | 6 and 10 weeks
  Overall patients status measured by the Patient Global Impression of Change (PGIC)
Change from baseline of the Social and Occupational Functioning Assessment Scale | 6 and 10 weeks
  Change from baseline of the Social and Occupational Functioning Assessment Scale (SOFAS)
Change from baseline of the Pittsburgh Sleep Quality Index | 6 and 10 weeks
  Change from baseline of the Pittsburgh Sleep Quality Index (PSQI)
Change from baseline of symptoms of PTSD and complex PTSD according to ICD-11 assessed with the International Trauma Questionnaire | 6 and 10 weeks
  Change from baseline of symptoms of PTSD and complex PTSD according to ICD-11 assessed with the International Trauma Questionnaire (ITQ)
Change from baseline of THC withdraw symptoms assessed with the Marijuana Withdrawal Checklist | 6 and 10 weeks and Follow- Up Visit 9
  Change from baseline of THC withdraw symptoms assessed with the Marijuana Withdrawal Checklist (MWC)
Responder analysis: proportion of patients showing improvement in nightmares | 10 weeks
  Responder analysis: proportion of patients showing improvement in nightmares (change from baseline) defined as decrease of CAPS-IV B2 ≥50% assessed at the end of treatment
Remitter analysis: proportion of patients showing full remission of nightmares | 10 weeks
  Remitter analysis: proportion of patients showing full remission of nightmares defined as CAPS-IV B2 = 0, assessed at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Roepke, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (4):
- Germany (4):
  - Berlin St. Hedwig, Berlin
  - Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin, Klinik für Psychiatrie und Psychotherapie, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Zentralinstitut für Seelische Gesundheit Mannheim, Mannheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roepke S, Schoofs N, Priebe K, Wulfing F, Schmahl C, Rohle R, Zahringer J, Lotter T, Otte C, Koglin S. Treating nightmares in posttraumatic stress disorder with dronabinol: study protocol of a multicenter randomized controlled study (THC PTSD-trial). BMC Psychiatry. 2023 May 5;23(1):319. doi: 10.1186/s12888-023-04818-5. PMID 37147642